CLINICAL TRIAL: NCT00350974
Title: Determination of Asymmetrical Dimethylarginine (ADMA) Accumulation in End Stage Renal Disease
Brief Title: ADMA Levels in End-Stage Renal Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Principal Investigator, Crystal A. Gadegbeku, Associate Professor of Internal Medicine, Nephrology, University of Michigan
Other Study IDs: HUM00004194
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Chronic Kidney Disease; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- End-stage Renal Disease: on maintenance hemodialysis 3 x per week for more than 12 months
- No kidney disease: eGFR greater than 60 ml/Min
- Hypertensive group: Blood pressure greater than 130/80

SUMMARY:
Asymmetric dimethylarginine, ADMA, in plasma, is significantly elevated in patients with renal disease and associated with cardiovascular morbidity and mortality. We found that whole blood (WB) possesses the metabolic pathways required for both the generation and elimination of ADMA and we have developed ex vivo methods to assess the WB accumulation of ADMA in humans. The over-arching hypothesis is that dysregulation of ADMA metabolic pathways leads to greater ADMA whole blood content and greater capacity to accumulate ADMA, which 1) is not reflected by plasma levels and 2) is a better predictor of cardiovascular outcome than plasma levels in end-stage renal disease (ESRD). The following specific aims will be pursued to characterize whole blood ADMA in ESRD:

1. Compare and contrast baseline free plasma ADMA and total whole blood (free plus protein-incorporated) ADMA concentrations in ESRD patients, matched hypertensive controls and a normal population.
2. Determine the capacity of WB to accumulate (the net balance of generation and elimination) ADMA in ESRD patients, matched hypertensive controls and a normal population.

We will use state-of-the-art, high performance liquid chromatography techniques to measure ADMA levels in plasma and whole blood. Samples for ADMA measurements will be obtained from subjects with end-stage renal disease immediately before their dialysis treatments. Samples will also be obtained from volunteers without kidney disease. This group will be matched to the end-stage renal volunteers by age, gender and ethnicity. These volunteers will also be matched for the presence of hypertension and diabetes. The third group will consist of a normal population to measure the normal levels of ADMA and compare to the other two groups.

There is growing evidence to support a pathological role of ADMA in humans. These experiments will enhance our understanding of how ADMA is processed in the human body and how it is associated with kidney disease. Potentially, these results will lay the groundwork for new insights into the link between ADMA and the high cardiovascular disease burden in patients with kidney disease.

ELIGIBILITY:
Inclusion

Group 1:

* are now 18 years of age or older, with end-stage renal disease (ESRD)
* have been on maintenance hemodialysis therapy three times/week for more then 12 months

Group 2 criteria:

* are now 18 years of age or older
* can be matched to a volunteer in Group 1 for age, gender, race, blood pressure and diabetes history
* have an eGFR greater then 60 ml/min (This is a value based on a laboratory blood test that shows how well your kidneys work.)

Group 3 criteria:

* are now 18 years of age or older
* have blood pressure less than 130/80 when you are not taking blood pressure medication
* normal kidney function

Exclusion

* are less then 18 years of age
* are pregnant or breast feeding
* unable or unwilling to provide informed consent
* are currently in another study
* have a hemoglobin (substance in red blood cells that carries oxygen) level that is less than 8 mg/dl
* have an untreated infection that won't go away
* require admission to the hospital
* have a history of hemolytic diseases (e.g. sickle cell disease)
* appear unlikely or unable to participate in the required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups: 16 healthy control subjects (CO), 18 patients with ESRD and 18 matched hypertensive patients with normal renal function (HTN).
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2006-07; Primary Completion 2007-03-08 (Actual); Study Completion 2007-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal A Gadegbeku, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States